CLINICAL TRIAL: NCT02098148
Title: A RANDOMIZED PLACEBO-CONTROLLED CROSSOVER TRIAL OF LOW-DOSE XENON FOR THE TREATMENT OF OBSESSIVE-COMPULSIVE DISORDER
Brief Title: Trial of Low-Dose Xenon For The Treatment Of Obsessive-Compulsive Disorder
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Withdrawn. Unable to set up appropriate infrastructure to support study.
Sponsor: Mclean Hospital (Other)
Responsible Party: Principal Investigator, Brian P. Brennan, MD, M.D., Mclean Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2013P001349
Record Dates: First submitted 2014-01-10; First posted 2014-03-27 (Estimated); Last update posted 2014-03-27 (Estimated); Status verified 2014-03

CONDITIONS: Obsessive-Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Xenon

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Xenon/Placebo (Experimental): Participants in this group will receive three treatments of 25% xenon followed by 3 treatments of placebo (room air).
  Interventions: Drug: Xenon; Drug: Placebo
- Placebo/Xenon (Experimental): Participants in this group will receive three treatments of placebo (room air) followed by three treatments of 25% xenon.
  Interventions: Drug: Xenon; Drug: Placebo

INTERVENTIONS:
Drug: Xenon
Drug: Placebo

SUMMARY:
The primary purpose of this study is to investigate whether administration of xenon reduces symptoms of Obsessive-Compulsive Disorder (OCD). Xenon is a naturally occurring gas that has been used in clinical settings both as a general anesthetic agent and as a contrast agent for computed tomography (CT) scans. Investigators believe that xenon may be effective in reducing symptoms of OCD due to its ability to reduce the activity of a specific brain chemical called glutamate, which has been shown to be abnormal in the brains of people with OCD.

It is important to understand that this study uses a placebo, or inactive, treatment. In this study, the placebo treatment is inhalation of room air (instead of xenon). All participants will receive both xenon and placebo treatments at some point over the course of the study. However, neither the participants nor the study investigators will know which treatment you are receiving.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female age ≥ 18 and ≤ 55
2. Meets DSM-IV criteria for OCD as primary presenting disorder
3. Score of ≥ 18 on the Y-BOCS at screening (Visit 1).

Exclusion Criteria:

1. Unwillingness or inability to provide written informed consent.
2. Lifetime history of schizophrenia or autism spectrum disorder
3. Diagnostic and Statistical Manual IV (DSM-IV) diagnosis of alcohol or substance dependence, with the exception of nicotine dependence, within three months prior to screening
4. Clinically significant medical disease including, but not limited to, pulmonary, cardiac (including uncontrolled hypertension), hepatic, renal, or endocrine disorders, which would increase the risk to the participant or interfere with interpretation of results as judged by the principal investigator.
5. Clinically significant neurologic disease including, but not limited to, seizure disorder, neurodegenerative diseases, and history of traumatic brain injury that would increase the risk to the participant or interfere with interpretation of results as judged by the principal investigator.
6. Female participants with a positive urine pregnancy test at screening
7. Pregnancy. Females of childbearing potential must be using an effective contraceptive method (e.g., abstinence, prescription oral contraceptives, contraceptive injections, double-barrier method, male partner sterilization).
8. Any screening laboratory abnormality deemed clinically significant by the investigator

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2013-11; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Decrease in OCD Symptoms | Baseline to Week 5
  Xenon is associated with a decrease in OCD symptoms as measured by the Yale-Brown Obsessive-Compulsive Scale (Y-BOCS) at completion of three treatments when compared to placebo (room air).

SECONDARY OUTCOMES:
Decrease in Depressive Symptoms | Baseline to Week 5
  Xenon is associated with a decrease in depressive symptoms as measured by the Montgomery-Asberg Depression Rating Scale (MADRS) at completion of three treatments when compared to placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Brian P Brennan, M.D., Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States